CLINICAL TRIAL: NCT04022265
Title: Bone Healing at Implants Installed in Sites Prepared Either With a Sonic Device or Drills. A Split-mouth Histomorphometric Randomized Controlled Trial
Brief Title: Bone Healing at Implants Installed in Sites Prepared Either With a Sonic Device or Drills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARDEC Academy (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: protocol #05-2014
Record Dates: First submitted 2019-07-11; First posted 2019-07-17 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Prostheses and Implants

STUDY DESIGN:
Intervention Model Description: Clinical Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Each patient will receive two mini-implants, installed in recipient sites prepared in the distal segments of the maxilla either with a sonic device or drills. The two recipient sites will be selected prior the surgery, while the type of site preparation will be randomly decided. A researcher, neither involved in the selection of the patients nor in the surgical and prosthetic treatment, carried out electronically the randomization (randomization.com). Sealed opaque envelopes will be prepared and opened at the time of surgery and they will report the position of the sonic sites so that the surgeon will be masked about site preparation type until the surgery. The site will be indicated as mesial or distal position if the two sites will be located in the same quadrant of the maxilla, or as right or left if they will be located in opposite quadrants of the maxilla.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Site -Drill site (Active Comparator): The control sites (Drills) will be prepared with a lanceolate drill (FS 230, Sweden / Martina), with a maximum diameter of 2.3 mm,
  Interventions: Device: implant placement
- Test site -sonic site (Experimental): test sites will be prepared with conical diamond inserts of increasing diameter (SFS99.000.014 to SFS99.000.024, Komet-Brasseler-GmbH, Germany) mounted on a sonic-air surgical instrument
  Interventions: Device: implant placement

INTERVENTIONS:
Device: implant placement — Full-thickness muco-periosteal flaps will be elevated, and the alveolar bone exposed to prepare the bed for the implant installation
  Other Names: implant surgery, prosthesis

SUMMARY:
The purpose was to evaluate histomorphometrically the early healing at implants installed in sites prepared with either a sonic device or conventional drills.

DETAILED DESCRIPTION:
Sixteen volunteer patients will be recruited. Two titanium mini-implants will be installed in the distal segments of the maxilla in recipient sites prepared with either a sonic device or conventional drills. Biopsies containing the mini-implants will be retrieved after 2 weeks in eight patients, and after 6 weeks in the other eight patients. Histomorphometric analyses will be performed

ELIGIBILITY:
Inclusion Criteria:

* presence of an edentulous atrophic zone in the posterior segment of the maxilla
* height of the sinus floor ≥10 mm
* ≥ 25 years of age;
* smoking ≤10 cigarettes per day
* good general health
* no contraindication for oral surgical procedures
* not being pregnant.

Exclusion Criteria:

* presence of systemic disorders
* chemotherapy or radiotherapy
* smokers >10 cigarettes per day
* previous bone augmentation procedures in the same region.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
New bone in contact with the implant surface | After 2 weeks to evaluate the healing prior to load with a prosthesis
  The percentages of new bone in contact with the implant surface will be evaluated in the histomorphometric analysis
New bone in contact with the implant surface | After 6 weeks, to evaluate the healing prior to load with a prosthesis
  The percentages of new bone in contact with the implant surface will be evaluated in the histomorphometric analysis

SECONDARY OUTCOMES:
The percentage of total mineralized bone in contact with the implant surface. | After 2 weeks to evaluate the healing prior to load with a prosthesis
  The percentages of new bone in contact with the implant surface will be evaluated in the histomorphometric analysis
The percentage of total mineralized bone in contact with the implant surface. | After 6 weeks to evaluate the healing prior to load with a prosthesis
  The percentages of new bone in contact with the implant surface will be evaluated in the histomorphometric analysis

OTHER OUTCOMES:
pre-existing (old) bone, soft tissues (marrow spaces, Haversian canals, BMUs canals), bone debris/ clot remnants, and vessels | After 2 weeks to evaluate the early haling prior to load with a prosthesis
  The percentages of pre-existing (old) bone, soft tissues (marrow spaces, Haversian canals, BMUs canals), bone debris/ clot remnants and vessels in contact with the implant surface will be evaluated in the histomorphometric analysis.
pre-existing (old) bone, soft tissues (marrow spaces, Haversian canals, BMUs canals), bone debris/ clot remnants, and vessels | After 6 weeks to evaluate the early haling prior to load with a prosthesis
  The percentages of pre-existing (old) bone, soft tissues (marrow spaces, Haversian canals, BMUs canals), bone debris/ clot remnants and vessels in contact with the implant surface will be evaluated in the histomorphometric analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Colombia, Cartagena, Cartagena, Colombia

IPD SHARING:
Plan to Share IPD: No
Will be shared after publication

REFERENCES:
- [Result] Atieh MA, Alsabeeha NHM, Tawse-Smith A, Duncan WJ. Piezoelectric versus conventional implant site preparation: A systematic review and meta-analysis. Clin Implant Dent Relat Res. 2018 Apr;20(2):261-270. doi: 10.1111/cid.12555. Epub 2017 Nov 16. PMID 29148161
- [Result] Bengazi F, Lang NP, Canciani E, Vigano P, Velez JU, Botticelli D. Osseointegration of implants with dendrimers surface characteristics installed conventionally or with Piezosurgery(R). A comparative study in the dog. Clin Oral Implants Res. 2014 Jan;25(1):10-5. doi: 10.1111/clr.12082. Epub 2012 Dec 12. PMID 23231427
- [Result] Vigano P, Botticelli D, Salata LA, Schweikert MT, Urbizo Velez J, Lang NP. Healing at implant sites prepared conventionally or by means of Sonosurgery (R). An experimental study in dogs. Clin Oral Implants Res. 2015 Apr;26(4):377-382. doi: 10.1111/clr.12348. Epub 2014 Feb 13. PMID 24524198
- [Result] Maurer P, Kriwalsky MS, Block Veras R, Vogel J, Syrowatka F, Heiss C. Micromorphometrical analysis of conventional osteotomy techniques and ultrasonic osteotomy at the rabbit skull. Clin Oral Implants Res. 2008 Jun;19(6):570-5. doi: 10.1111/j.1600-0501.2007.01516.x. PMID 18474063
- [Result] Schaeren S, Jaquiery C, Heberer M, Tolnay M, Vercellotti T, Martin I. Assessment of nerve damage using a novel ultrasonic device for bone cutting. J Oral Maxillofac Surg. 2008 Mar;66(3):593-6. doi: 10.1016/j.joms.2007.03.025. No abstract available. PMID 18280402
- [Result] Stacchi C, Berton F, Turco G, Franco M, Navarra CO, Andolsek F, Maglione M, Di Lenarda R. Micromorphometric analysis of bone blocks harvested with eight different ultrasonic and sonic devices for osseous surgery. J Craniomaxillofac Surg. 2016 Sep;44(9):1143-51. doi: 10.1016/j.jcms.2016.04.024. Epub 2016 Apr 22. PMID 27527676
- [Result] Amghar-Maach S, Sanchez-Torres A, Camps-Font O, Gay-Escoda C. Piezoelectric surgery versus conventional drilling for implant site preparation: a meta-analysis. J Prosthodont Res. 2018 Oct;62(4):391-396. doi: 10.1016/j.jpor.2018.04.004. Epub 2018 May 26. PMID 29843978
- [Result] Sendyk DI, de Oliveira NK, Pannuti CM, da Graca Naclerio-Homem M, Wennerberg A, Deboni MCZ. Conventional Drilling Versus Piezosurgery for Implant Site Preparation: A Meta-Analysis. J Oral Implantol. 2018 Oct;44(5):400-405. doi: 10.1563/aaid-joi-D-17-00091. Epub 2018 Mar 27. PMID 29583059
- [Result] Stacchi C, Vercellotti T, Torelli L, Furlan F, Di Lenarda R. Changes in implant stability using different site preparation techniques: twist drills versus piezosurgery. A single-blinded, randomized, controlled clinical trial. Clin Implant Dent Relat Res. 2013 Apr;15(2):188-97. doi: 10.1111/j.1708-8208.2011.00341.x. Epub 2011 Apr 19. PMID 21682844
- [Result] Preti G, Martinasso G, Peirone B, Navone R, Manzella C, Muzio G, Russo C, Canuto RA, Schierano G. Cytokines and growth factors involved in the osseointegration of oral titanium implants positioned using piezoelectric bone surgery versus a drill technique: a pilot study in minipigs. J Periodontol. 2007 Apr;78(4):716-22. doi: 10.1902/jop.2007.060285. PMID 17397320
- [Result] Geminiani A, Papadimitriou DE, Ercoli C. Maxillary sinus augmentation with a sonic handpiece for the osteotomy of the lateral window: a clinical report. J Prosthet Dent. 2011 Nov;106(5):279-83. doi: 10.1016/S0022-3913(11)00143-0. PMID 22024176
- [Result] Geminiani A, Weitz DS, Ercoli C, Feng C, Caton JG, Papadimitriou DE. A comparative study of the incidence of Schneiderian membrane perforations during maxillary sinus augmentation with a sonic oscillating handpiece versus a conventional turbine handpiece. Clin Implant Dent Relat Res. 2015 Apr;17(2):327-34. doi: 10.1111/cid.12110. Epub 2013 Jul 9. PMID 23837594
- [Result] Papadimitriou DE, Geminiani A, Zahavi T, Ercoli C. Sonosurgery for atraumatic tooth extraction: a clinical report. J Prosthet Dent. 2012 Dec;108(6):339-43. doi: 10.1016/S0022-3913(12)00169-2. PMID 23217465
- [Result] Agabiti I, Cappare P, Gherlone EF, Mortellaro C, Bruschi GB, Crespi R. New surgical technique and distraction osteogenesis for ankylosed dental movement. J Craniofac Surg. 2014 May;25(3):828-30. doi: 10.1097/SCS.0000000000000737. PMID 24777021
- [Result] Agabiti I, Bernardello F, Nevins M, Wang HL. Impacted canine extraction by ridge expansion using air scaler surgical instruments: a case report. Int J Periodontics Restorative Dent. 2014 Sep-Oct;34(5):681-7. doi: 10.11607/prd.1884. PMID 25171039
- [Result] Agabiti I, Botticelli D. Two-Stage Ridge Split at Narrow Alveolar Mandibular Bone Ridges. J Oral Maxillofac Surg. 2017 Oct;75(10):2115.e1-2115.e12. doi: 10.1016/j.joms.2017.05.015. Epub 2017 May 24. PMID 28623685
- [Result] Heinemann F, Hasan I, Kunert-Keil C, Gotz W, Gedrange T, Spassov A, Schweppe J, Gredes T. Experimental and histological investigations of the bone using two different oscillating osteotomy techniques compared with conventional rotary osteotomy. Ann Anat. 2012 Mar 20;194(2):165-70. doi: 10.1016/j.aanat.2011.10.005. Epub 2011 Oct 17. PMID 22056295
- [Result] Caneva M, Lang NP, Calvo Guirado JL, Spriano S, Iezzi G, Botticelli D. Bone healing at bicortically installed implants with different surface configurations. An experimental study in rabbits. Clin Oral Implants Res. 2015 Mar;26(3):293-9. doi: 10.1111/clr.12475. Epub 2014 Sep 15. PMID 25220835
- [Result] Ferri M, Lang NP, Angarita Alfonso EE, Bedoya Quintero ID, Burgos EM, Botticelli D. Use of sonic instruments for implant biopsy retrieval. Clin Oral Implants Res. 2015 Nov;26(11):1237-43. doi: 10.1111/clr.12466. Epub 2014 Aug 11. PMID 25109369
- [Result] Botticelli D, Lang NP. Dynamics of osseointegration in various human and animal models - a comparative analysis. Clin Oral Implants Res. 2017 Jun;28(6):742-748. doi: 10.1111/clr.12872. Epub 2016 May 23. PMID 27214566

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT04022265/Prot_SAP_000.pdf